CLINICAL TRIAL: NCT02671409
Title: Translational Study of the Effects of Neural Mobilization in Patients With Lomboisquiatalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, marucia chacur, PHD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2 44079115.1.1001.5511
Record Dates: First submitted 2016-01-29; First posted 2016-02-02 (Estimated); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Low Back Pain, Mechanical; Pain; Neuropathic Pain
MeSH Terms: conditions — Low Back Pain; Pain; Neuralgia | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (Placebo Comparator): The exercise program will be drawn from the recommendations of the American College of Physicians and the American Pain Society for the treatment of low back pain. The exercise protocol consist of: Strengthening the abdominal muscles and erector spinae: will be three sets of 15 repetitions for each exercise with rest time between 2 minutes series; - Proprioceptive Neuromuscular Facilitation (PNF). The PNF technique will be the contract-relax the hamstrings by 6/2. Stretching the erector muscles of the spine, iliopsos, hamstrings, quadriceps and sural triceps: will be three three repetitions, with 30 seconds support time each stretch and rest time between sets 1 minute.
  Interventions: Other: Neural Mobilization (exercise)
- MOB Group (Experimental): Initially patients will be informed about the procedures. After the guidelines, the hip and knee are palpated to start the joint angles. Then, the knee joint is positioned in extension and remained so throughout the treatment. In addition, the hip joint is bent until the moment that will be perceived a minimum strength of the muscles of the posterior region of thigh and leg (discarding muscle stretching). Neural mobilization is started at the time when the ankle joint will be manipulated in dorsiflexion at a frequency of approximately 20 oscillations per minute, with a pause of 25 seconds of rest. In the last two minutes of therapy, we will include cervical flexion, in order to intend the neuraxis, keeping artuculares amplitudes.
  Interventions: Other: Neural Mobilization (exercise)

INTERVENTIONS:
Other: Neural Mobilization (exercise) — Initially patients will be informed about the procedures. After the guidelines, the hip and knee are palpated to start the joint angles. Then, the knee joint is positioned in extension and remained so throughout the treatment. In addition, the hip joint is bent until the moment that will be perceived a minimum strength of the muscles of the posterior region of thigh and leg (discarding muscle stretching). Neural mobilization is started at the time when the ankle joint will be manipulated in dorsiflexion at a frequency of approximately 20 oscillations per minute, with a pause of 25 seconds of rest. In the last two minutes of therapy, we will include cervical flexion, in order to intend the neuraxis, keeping artuculares amplitudes.

SUMMARY:
The spinal nerve injury in humans often results in neuropathic pain characterized by spontaneous burning pain accompanied by allodynia and hyperalgesia. In this sense, lomboisquiatalgia is a neuropathy that is characterized by narrowing the intervertebral foramen of the lumbar vertebrae, leading a lumbar chronic pain which irradiate to a lower limb, being a clinical condition of difficult treatment. Neural Mobilization is a noninvasive technique used by physiotherapists. The technique aims to restore mobility and elasticity of the peripheral nervous system by tenses which are imposed on the roots, nerves, spinal cord and their respective meninges. This technique has been standardized in basic research and has shown promising results. However, clinically, this technique lacks randomized, controlled and double blind studies. Therefore, the investigators have to evaluate the effects of Neural Mobilization technique in patients with lomboisquiatalgia. In this study the investigators will treat patients three times a week, with ten minute treatment time per session, with 25 oscillations per minute for ten sessions. Many tools will be used to assess the effects of the protocol applied, for example: evaluation sheet, visual analogue scale (VAS), quality of life assessment - WHOQOL-bref questionnaire of Roland Morris disability, oswestry index on disability (version 2.0), enzyme-linked immunosorbent assays for the measurement of cytokines in the blood tissue. In this way, the investigators can contribute and understand the mechanisms involved in the rehabilitation process.

DETAILED DESCRIPTION:
Translational study of the effects of Neural Mobilization in patients with lomboisquiatalgia

The spinal nerve injury in humans often results in neuropathic pain characterized by spontaneous burning pain accompanied by allodynia and hyperalgesia [1]. These signs and symptoms occur in the continuous presence of ectopic focus of the afferent peripheral nervous system (peripheral sensitization) to the central nervous system (CNS) (central sensitization). After the traumatic experience both peripheral sensitization and central sensitization contributes to the appearance of poorly adaptive responses in the spinal cord as well as in the brain, contributing to chronicity and maintenance of neuropathic pain [2, 3]. The pain-induced neuropathy is currently being associated with the involvement of glial cells located in the spinal cord [4, 5]. Glial cells synthesize several substances, many of which are also released by nociceptive neurons that modulate the pain response, among which we can mention prostaglandins, glutamate, arachidonic acid, nitric oxide and cytokines pro inflammatory [6-9]. Pro-inflammatory cytokines appear to be involved in hyperalgesia and mechanical allodynia arising from nerve injury due to compression. Many studies have demonstrated that in models of peripheral nerve trunks ischemia, in rats, occurs an increase in pro-inflammatory cytokines that may be related to myelin damage and edema [10, 11]. Furthermore, studies using nerve compression model, increased identified interleukins (IL-6 or TNF) in rats with allodynia [12]. In this sense, the interleukins (IL) are proteins produced by T groups and many of these cells are involved in IL activation of lymphocytes, each of which has its effect on IL specific groups of cells expressing specific receptors which are identified by numbers: IL-1, IL4, IL-6, IL-10 [13]. Kraychete et. al. (2009), analyzed by means of blood samples the levels of pro-inflammatory cytokines in the plasma of patients with and without neuropathic pain, and found that patients with neuropathies had higher levels of these cytokines [14]. Kukkar et. al. (2012), a model of neuropathic pain (CCI) observed an increase of TNF-α level in the sciatic nerve after treatment with aliskiren (an anti-hipertensive drug) and a decrease in TNF-α with consequent improvement in nociception [15].

In clinical practice, has been extensively reported that neuropathic pain is difficult to treat due to inadequate understanding of the cellular and molecular mechanisms involved in the development and maintenance of this kind of pain [16, 17]. The therapeutic options for the control of neuropathic pain have increased in recent years [18]. However, responses to treatments is still not satisfactory. The neurosurgical treatments include pharmacological treatments, such as antidepressants, anticonvulsants, gabapentin, carbamazepine, systemic administration of local anesthetics, topical agents, narcotic analgesics and non-narcotic antiarrhythmics [17, 18]. Still, as a complementary non-invasive and non-pharmacological treatment, we find in the literature, the use of therapeutic resources for rehabilitation, depending on the kinf of injury. In this context, Neural Mobilization techniques have shown excellent prognosis in patients with differents kind of pain, besides other advantages, such as low operating cost, easy to use and no adverse effects [19]. Neural Mobilization is a noninvasive technique used by physiotherapists, this technique aims is, to restore mobility and elasticity of the peripheral nervous system by strains imposed on nerve trunks, roots, nerves, spinal cord and their wraps, the meninges due to the imposition of movements and joint angles [20].

Currently, the technique has been used as a method of evaluation and treatment of several diseases that affect the central nervous system (such as Stroke) or peripheral (herniated discs or nerve impingement) and structures such as, the muscles due to the existing integration between the musculoskeletal system and the nervous system [19, 21-23]. The healthy relationship, away from injuries, between peripheral nerves and locomotor system with respect to their tissue interfaces allows individuals to move from free and without pain [24]. Research by Dworkin et al., (2007) points out that the Neural mobilization is effective in conditions of musculoskeletal injuries to functional and pathological diagnosis [21]. However, the authors mention that for each musculoskeletal condition a kind of neural mobilization should be performed. Also depending on the clinical condition of the patient other therapies may be included in treatment plan. Our group has been studying last six years, and standardizing the technique Neural Mobilization (MOB) in rats. Encouraging results were found using our treatment protocol. We demonstrated that the MOB reduced nociceptive frame, through the involvement of opioid receptors in the central nervous system (PAG) and peripheral (DRG), involvement of substance P, TRPV 1, NGF, PO (protein zero), intense regeneration process in sciatic nerve and, exponential increase in muscle strength [25-28,34]. Thus, we believe that Neural Mobilization technique, through basic research, appears to be effective in the antinociceptive process.

EXPECTED RESULTS:

Is consensus that therapeutic alternatives for the treatment of neuropathic pain are needed. Physical therapy has been shown by Neural Mobilization technique is efetive in pain control. This project becomes important because of the lack of consistent controlled, randomized and double blind, demonstrating the benefits effect of Neural Mobilization technique in patients with neuropathic pain. The lomboisquiatalgia is characterized by narrowing of the intervertebral foramen of the lumbar vertebrae and spinal nerve projection site. It is a clinical complication difficult to diagnose and very easy to be confused with herniated disc, piriformis syndrome or even osteoarthritis disc. The isquiatalgia is induced by nerve root compression (local projection roots which form the sciatic nerve between L3 and L4 and L5 and S1), most often caused by a protrusion of nucleus pulposus by virtue of disruption of the fibrous rings symphysis intervertebral [30]. Neural mobilization technique is able to induces an antinociceptive effect in model of cronic pain, reason it is an important clinical tool in the treatment of patients with neuropathic pain [28, 20, 31]. Thus, we believe that we need to perform, randomize, control the frequently sessions and time of treatment to bring from basic research to now to the clinic in order to better understand the mechanism involved in this kind of pain. In this way, we can contribute effectively and understand the mechanisms involved in the rehabilitation process of these patients, correlating with improvement in pain and consequent improvement of life of patients.

AINS

Evaluate the effects of Neural Mobilization technique on the quality of life, biochemical changes in patients with lomboisquiatalgia using:

* Check the immediate effect of neural mobilization technique on pain of patients with lomboisquiatalgia through pain scale;
* Check and analysis if Neural mobilization technique increase the functional of patients with lomboisquiatalgia;
* Examine the impact of treatment with Neural Mobilization in pro- and anti inflammatory citokynes (IL-1β, IL-6, IL-10, TNFa and fractalquina) through the analysis of patients blood tissue;
* Check possible adverse effects of Neural Mobilization technique in patients with lomboisquiatalgia.

SCIENTIFIC AND TECHNOLOGICAL CHALLENGES AND THE MEANS AND METHODS TO OVERCOME THEM

* Study and ethics of design: will be a randomized, controlled, double-blind, in accordance with the ethical standards of the Declaration of Helsinki, as approved by the Ethics Committee in Research with Human Subjects at the University Nove , São Paulo, SP, Brazil (2 44079115.1.1001.5511).
* Participants: Subjects will be recruited from the Integrated Health Clinic at the University Nove in Sao Paulo / SP, even through phone contact, e-mail and letters to orthopedic doctors, clinicians and neurologists. Potentially eligible subjects will be invited for an interview and a screening procedure performed by a physiotherapist. After eligibility, subjects will sign the Term of Free and Clear (TCLE), according to Resolution 196/96 of the National Health Council, confirming the participation in the survey.
* Calculation of the sample: The sample size was calculated based on the Analog Scale pain, which was considered the primary end point. To this end, the variance reported in a study by Murphy et al., 2006, whose objective was to evaluate the Neural mobilization as a technique for the treatment of lumbar spinal stenosis. Considering the mean and standard deviation of the pre- intervention and post-intervention this study, with an alpha value ( α ) of 0.05 and 90% power test, it was determined that 40 subjects were required , It is 20 for each experimental group and 20 for each control group [32].

Evaluation of outcomes

* Visual Analogue Scale: The primary outcome of interest will be assessed by Visual Analogue Scale (VAS). The VAS is to assist in the assessment of pain intensity in the participant.
* Questionnaire WHOQOL-BREF: The WHOQOL-bref questionnaire is a specific questionnaire, short and quick application, developed by the World Health Organization (WHO) in order to standardize the assessment of quality of life.
* Disability Questionnaire Roland Morris - RMDQ: Roland and Morris developed in 1983 a questionnaire to assess functional disability of patients with low back pain.
* Oswestry Disability Index (ODQ - version 2.0): The Oswestry disability Index (Oswestry Low Back Pain Disability Questionnaire (ODQ) aims to assess dysfunction in individuals with low back pain by analyzing the activities of daily living.
* Enzyme-linked immunosorbent assays for the measurement of cytokines: To assess the impact of Neural Mobilization technical front of interleukin pro- and anti-inflammatory collecting blood tissue will be necessary (for blood collection will follow the manual techniques for collection ministry of Health of the blood [33] of each patient to the enzyme immunoassays for each specific cytokine). Will be made two blood collections, the original measure (the first session) and after the last session (tenth session) treatment. The blood tissue will initially be stored after collection and centrifuged for 20 minutes at 3000 rpm. For dosage fractalkine, cytokines (IL-1β, IL-6 and IL-10 and TNF-α) specific reagents will be used in Milliplex®TM Map Kit (Millipore Corporation, Darmstadt- Germany) according to the protocol specified by the manufacturer.

REFERENCES - I excuse references because have limit of characters

ELIGIBILITY:
Inclusion Criteria: Selected will be subject to meeting the following criteria: chronic low back pain radiating to the leg for more than three months from the narrowing of the intervertebral foramen of the lumbar vertebrae (lomboisquiatalgia), ie for more than 12 weeks; age ≥ 20 years; score ≥ 4 on analog pain scale (VAS); DN4 ≥ 4 on scale; both genders; positive for the following special tests: Slump-Test, the straight leg raising test, Lasègue Test, Rise Of Opposite Leg and Sign of Arc or Bowstring-Sign rope; score ≥ 4 on the Roland Morris Disability Questionnaire (RMDQ); ≥ moderate dysfunction in Oswestry Low Back Pain Disability Questionnaire.

Exclusion Criteria: Will be excluded from study subjects with the presence aged over 35 years, acute lumbar pain; recent history of violent trauma; spondylolisthesis or fibromyalgia; previous surgery column, any sequel that causes limitation in the lower limb range of motion (joint deformity), subjects suffering precaution for Neural Mobilization or cortical stimulation transmagnética as pacemaker, metal plates, screws, neurological disorders; systemic disease, immunosuppression, cancer patients, psychological disorders, cognitive disorders and failure, any kind of pain in other regions is not characteristic of lomboisquiatalgia and lack of cooperation or cognitive capacity to perform clinical procedures and pregnant women. The subjects will be kept blind to the treatment allocation. Researchers involved in the application of techniques will be kept blind throughout the development and analysis of the study.

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2016-10; Primary Completion 2019-03 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Pain: Visual Analog Scale | 1 month
  VAS - Visual Analog Scale

SECONDARY OUTCOMES:
Quality of life: Questionnaire WHOQOL-bref | 1 month
  Questionnaire WHOQOL-bref

OTHER OUTCOMES:
Disability functional: Questionnaire Roland Morris - RMDQ | 1 month
  Questionnaire Roland Morris - RMDQ
Assess dysfunction in individuals with low back pain by analyzing the activities of daily living: Oswestry Low Back Pain Disability Questionnaire | 1 month
  Oswestry Low Back Pain Disability Questionnaire (ODQ)
Cytokine assay: immunohistochemistry - Milliplex®TM Map | 1 month
  Immunohistochemistry - Milliplex®TM Map (Millipore Corporation, Darmstadt- Germany)

CONTACTS AND LOCATIONS:
Overall Officials: FABIO MARTINEZ DOS SANTOS, PHD, Principal Investigator — University of Sao Paulo; MARINA RAMOS, PT, Principal Investigator — University of Sao Paulo; MARUCIA CHACUR, PHD, Study Chair — University of Sao Paulo
Locations (1):
- University of Sao Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
semi-annual report

DOCUMENTS (2):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form: Study Protocol (2018-09-10): https://cdn.clinicaltrials.gov/large-docs/09/NCT02671409/Prot_SAP_ICF_000.pdf
  • Study Protocol: New protocol (2019-03-10): https://cdn.clinicaltrials.gov/large-docs/09/NCT02671409/Prot_001.pdf